CLINICAL TRIAL: NCT02514863
Title: Influence of Electrode Placement on Electrical Velocimetry Cardiac Output Measurements
Brief Title: Electrode Placement in Electrical Velocimetry
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2009-MA-electrodes
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing CMR: Assessment of hemodynamic function using:
  * CMR
  * EV with an inter-electrode gap (lower pair) of 5 cm
  * EV with an inter-electrode gap (lower pair) of 15 cm

SUMMARY:
Electrical velocimetry (EV) is one of the latest adaptions of impedance cardiography showing diverging results. With electrode position being a suspected factor influencing measurement accuracy or reproducibility for impedance cardiography in general, no data is currently available on altering the gap of the two lower electrodes in EV. Reference values were determined using the non-invasive gold-standard cardiac magnetic resonance imaging (CMR).

ELIGIBILITY:
Inclusion Criteria:

* indication for CMR

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing CMR
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
difference between CMR and EV cardiac output measurements | 45 minutes

SECONDARY OUTCOMES:
difference between two consecutive EV cardiac output measurements | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Mannheim, Mannheim, Germany